CLINICAL TRIAL: NCT04449315
Title: Outpatient Oncology Aromatherapy
Brief Title: Outpatient Oncology Aromatherapy for Symptom Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central DuPage Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CentralDuPage
Record Dates: First submitted 2020-06-12; First posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Anxiety; Nausea
MeSH Terms: conditions — Anxiety Disorders; Nausea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peppermint and Lavender Essential Oil (Experimental): Young Living Essential oil of Peppermint and Lavender will be used to patients who meet the inclusion criteria.
  Interventions: Other: Young Living Lavender Essential Oil

INTERVENTIONS:
Other: Young Living Lavender Essential Oil — For qualified patients one to two drops of hospital approved essential oil will be placed on a 4X4 gauze and will be offered to the patient during their infusion visit. This gauze will be placed in a sealable clear plastic bag and the patient will be instructed to use one sniff at a time.
  Other Names: Young Living Peppermint Essential Oil

SUMMARY:
The purpose of this research study is to determine whether using aromatherapy during chemotherapy infusion treatments in the outpatient Oncology setting promote relief of nausea and anxiety.

The objectives of this study are: 1. To promote relief of nausea using peppermint aromatherapy oil in an outpatient oncology setting. 2. To promote relief of anxiety using lavender aromatherapy oil in an outpatient oncology setting.

DETAILED DESCRIPTION:
Subject Selection: Every outpatient oncology patient experiencing nausea and/or anxiety during an infusion visit will be offered hospital-approved aromatherapy of Peppermint oil or Lavender oil. If patient says yes, then they will be selected for the study and infusion nurse will notify the study co-investigators or principal investigator. Informed consent will then be obtained by co-investigators or principal investigator of the study. The consents as well as the data collection tool sheets will be numbered without identifying patient's personal information. Peppermint oil aromatherapy and/or lavender oil aromatherapy will then be administered to consented patients.

Method of Subject Identification and Recruitment: Every outpatient oncology patient experiencing nausea and/or anxiety during an infusion visit will be offered hospital- approved aromatherapy of Peppermint oil or Lavender oil. If patient says yes, then they will be selected for the study and infusion nurse will notify the study co-investigators or principal investigator. Informed consent will then be obtained by co-investigators or principal investigator of the study. The consents as well as the data collection tool sheets will be numbered without identifying patient's personal information. Peppermint oil aromatherapy and/or lavender oil aromatherapy will then be administered to consented patients.

ELIGIBILITY:
Inclusion Criteria:

All outpatient Oncology patients > 18 years of age Non pregnant Not cognitively impaired English speaking only Patients who report nausea and/or anxiety

Exclusion Criteria:

All outpatient oncology patients <18 years of age Pregnant Cognitively impaired Non-English Speaking Patients who do not report nausea and/or anxiety Patients with a known allergy to peppermint and/or lavender aromatherapy oil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Post Intervention Interview From | Immediately upon Completion of the patient's infusion
  After the patients' infusion they will be asked questions from this form

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine Mack, MSN, Principal Investigator — Central DuPage Hospital
Locations (1):
- Central DuPage, Winfield, Illinois, United States

IPD SHARING:
Plan to Share IPD: No